CLINICAL TRIAL: NCT00715884
Title: A Prospective, Single-Blind, Randomized, Multi-Center Study Comparing the CYPHER® ELITE™ to the CYPHER® Bx VELOCITY® Sirolimus-Eluting Stent Systems (ELITE).
Brief Title: Study Comparing the CYPHER® ELITE™ to the CYPHER® Bx VELOCITY® Sirolimus-Eluting Stent Systems
Acronym: ELITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P07-6330
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerosis
Keywords: Atherosclerosis; de novo native coronary lesion
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CYPHER® ELITE™ Sirolimus-Eluting Stent System.
  Interventions: Device: CYPHER® ELITE™ Sirolimus-Eluting Stent System
- 2 (Active Comparator): CYPHER® Bx VELOCITY® Sirolimus-eluting Stent System
  Interventions: Device: CYPHER® Bx VELOCITY® Sirolimus-eluting Stent System

INTERVENTIONS:
Device: CYPHER® ELITE™ Sirolimus-Eluting Stent System — Drug eluting stent
  Other Names: Cypher ELITE
  Arms: 1
Device: CYPHER® Bx VELOCITY® Sirolimus-eluting Stent System — Drug eluting stent
  Other Names: CYPHER Bx VELOCITY
  Arms: 2

SUMMARY:
The objective of this study is to show similar (non-inferior) safety and effectiveness between CYPHER® ELITE™ and CYPHER® Bx VELOCITY® Sirolimus-Eluting Stent Systems in a prospective, multi-center, randomized clinical study for the treatment of de novo native coronary lesions.

DETAILED DESCRIPTION:
A prospective, single-blind, randomized, multicenter, two arm study. The objective of this study is to show similar (non-inferior) safety and effectiveness between CYPHER® ELITE™ and CYPHER® Bx VELOCITY® Sirolimus-Eluting Stent Systems in a prospective, multi-center, randomized clinical study for the treatment of de novo native coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with de novo atherosclerotic CAD in 1 or 2 vessels;
* The subject must be >/= 18 years of age;
* Female of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment;
* Diagnosis of angina pectoris as defined by stable angina pectoris Canadian Cardiovascular Society Classification (Class I, II, III) OR non-ST segment elevation acute coronary syndrome (Braunwald Classification B&C) OR non-ST segment elevation myocardial infarction >/= 48 hours from the time of study index procedure OR asymptomatic subjects with a positive stress test;
* Treatment of </= two lesions in one or two major coronary arteries (1 target lesion in each of 2 vessels or 2 target lesions in 1 vessel);
* Target vessel diameter must be >/= 2.25mm and </= 4.0 in diameter (visual estimate);
* Target lesion stenosis is > 50% and < 100% (visual estimate);
* Target lesion length <30mm (for each target lesion(s)) with a total implanted stent length < 66mm. Additional stents can be used to treat dissections, etc,: however, these must be the same stent to which the subject has been randomized in the study.
* Subject or Legally Authorized Representative must provide written informed consent prior to the procedure using a form that is approved by the Institutional Review Board/Independent Ethics Committee.

Exclusion Criteria:

* ST Segment Elevation Myocardial Infarction (STEMI) within 30 days of the study index procedure;
* Unprotected left main coronary disease with >/= 50% stenosis;
* Total coronary occlusion or TIMI grade 0 or 1 in the target vessel;
* Angiographic evidence of thrombus within target lesion(s);
* Calcified target lesion(s) which cannot be, in the investigator's opinion, successfully pre-dilated;
* Bifurcation disease involving a side branch >/= 2 mm in diameter;
* Prior stent within 5 mm of target lesion(s);
* Ostial target lesion(s);
* Target lesion(s) within a coronary bypass graft (e.g., saphenous vein or arterial graft);
* Documented left ventricular ejection fraction </= 25%;
* Impaired renal function (creatinine > 250 μmol/L or > 2.5 mg/dl) at the time of treatment;
* Pretreatment with devices other than conventional balloon angioplasty;
* Significant angulation in the target vessel that, in the Investigator's opinion, may preclude stent delivery and deployment;
* Subject previously treated with brachytherapy;
* Recipient of heart transplant;
* Subject with a life expectancy less than 12 months;
* Known allergies to the following: aspirin, clopidogrel bisulfate and ticlopidine, heparin, stainless steel, contrast agent (that cannot be managed medically), or sirolimus that cannot be managed medically;
* Any significant medical condition which, in the Investigator's opinion, may interfere with the subject's optimal participation in the study;
* Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the study endpoints;
* In the Investigator's opinion, the lesion is not suitable for stenting;
* Known bleeding or hypercoagulable disorder;
* Known or suspected active infection at the time of the study procedures;
* Subject is known to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser;
* Subject has had major surgical or interventional procedures unrelated to this study within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2014-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Satler, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ELITE™: CYPHER® ELITE™ Sirolimus-Eluting Stent System.
- CYPHER®: CYPHER® Bx VELOCITY® Sirolimus-eluting Stent System
Period: Overall Study
Arm/Group | ELITE™ | CYPHER®
Started | 452 | 226
Completed | 444 | 225
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELITE™ | CYPHER® | Total
Number analyzed (Participants) | 452 | 226 | 678
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 137 | 389
  >=65 years | 200 | 89 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.5) | 62.2 (10.5) | 62.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 74 | 212
  Male | 314 | 152 | 466
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 4 | 25
  Not Hispanic or Latino | 421 | 218 | 639
  Unknown or Not Reported | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 452 | 226 | 678
Race [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 11 | 3 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 20 | 53
  White | 403 | 203 | 606
  Other | 3 | 0 | 3
Patients with History of Previous Percutaneous Coronary Intervention (PCI) [Number; unit: participants]
  History of Previous PCI | 145 | 69 | 214
  Without History of Previous PCI | 307 | 157 | 464
Patients with History of Previous Coronary Artery Bypass Graft (CABG) [Number; unit: participants]
  History of Previous CABG | 48 | 21 | 69
  Without History of Previous CABG | 404 | 205 | 609
Patients with Family History of Coronary Artery (CAD) [Number; unit: participants]
  Family History of Coronary Artery (CAD) | 255 | 137 | 392
  Without Family History of Coronary Artery (CAD) | 197 | 89 | 286
Patients with History of Hyperlipidemia [Number; unit: participants]
  History of Hyperlipidemia | 388 | 188 | 576
  Without History of Hyperlipidemia | 64 | 38 | 102
Patients with History of Hypertension [Number; unit: participants]
  History of Hypertension | 360 | 178 | 538
  Without History of Hypertension | 92 | 48 | 140
Patients with History of Diabetes Mellitus [Number; unit: participants]
  History of Diabetes Mellitus | 144 | 69 | 213
  Without History of Diabetes Mellitus | 308 | 157 | 465

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Target Lesion Failure (TLF)
Description: The primary endpoint for this study is the percentage of participants who experienced Target Lesion Failure (TLF) during the 12 months post-procedure. A TLF event is defined as clinically-driven target lesion revascularization, target vessel myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel at 12 months post-procedure.
Time Frame: 12-months post-procedure
Population: Event-specific adjusted intent to treat (ITT) population: All randomized participants excluding those with follow-up less than 330 days and without documented events during the 360 days post procedure
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 429 | 216
Percentage of participants | 5.36 | 2.78
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Sample sizes of 1,061 from the ELITE™ group and 531 from the CYPHER® group were planned to achieve 90 percent power at a 2.5 percent significance level using an one-sided equivalence test, assuming a 10 percent TLF rate in each group and the maximum allowable rate difference between the groups being 5 percent. The total sample size was increased to 1,770 patients to account for an approximately 90 percent compliance to clinical follow-up; Test type: Non-Inferiority or Equivalence — The null inferiority hypothesis was that the upper limit of the 95% confidence interval is equal or greater than the non-inferiority margin 5%. The alternative non-inferiority hypothesis for this study assumed that the upper limit of the 95% confidence interval would be less than the non-inferiority margin 5%; In the CYPHER® ELITE™ arm the TLF rate was 5.36% (23/429) compared with 2.78% (6/216) in the CYPHER® Bx VELOCITY® arm, a difference in rates of 2.58%, upper limit of 95% two sided confidence interval of 5.55%; Difference between TLF rates = 2.58, 95% CI 1-sided [upper limit 5.55]

2. Secondary Outcome: Percentage of Lesion Success
Description: Lesion success is defined as the attainment of < 50 percent residual stenosis (by Quantitative Coronary Angiography (QCA)) using any percutaneous method.
Time Frame: At procedure
Population: ITT: All randomized participants regardless whether they received the intervention
Measure: Number; unit: Percentage of success
Units Other Than Participants: Lesions
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 452 | 226
Number analyzed (Lesions) | 538 | 281
Percentage of success | 99.6 | 100.0
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.549, Fisher Exact; Difference between event rates = -0.4, 95% CI 2-sided [-1.3 to 1.0]

3. Secondary Outcome: Percentage of Device Success - Protocol Definition
Description: Device success is defined as achievement of a final residual diameter stenosis of <50 percent (by QCA), using the assigned device only. If QCA was not available, the visual estimate of diameter stenosis was used. Device success was based on the following two measurements. Protocol definition: Only protocol-defined study stents were included.
Time Frame: At procedure
Population: Intent to Treat population.
Measure: Number; unit: Percentage of success
Units Other Than Participants: Devices
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 452 | 226
Number analyzed (Devices) | 541 | 283
Percentage of success | 95.7 | 82.0
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p < .001, Fisher Exact; Difference between event rates = 13.8, 95% CI 2-sided [9.2 to 18.9]

4. Secondary Outcome: Percentage of Device Success - All CYPHER® Stents Included
Description: Device success is defined as achievement of a final residual diameter stenosis of <50 percent (by QCA), using the assigned device only. If QCA was not available, the visual estimate of diameter stenosis was used. Device success was based on the following two measurements. All CYPHER® Stents were included if the final residual stenosis was <50%. Non-study CYPHER® Stents were also included.
Time Frame: At procedure
Population: Intent to Treat population.
Measure: Number; unit: Percentage of success
Units Other Than Participants: Devices
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 452 | 226
Number analyzed (Devices) | 538 | 283
Percentage of success | 95.7 | 95.1
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.724, Fisher Exact; Difference between event rates = 0.7, 95% CI 2-sided [-2.2 to 4.2]

5. Secondary Outcome: Percentage of Participants Who Achieved Procedure Success
Description: Procedure success is defined as achievement of a final diameter stenosis of < 50 percent (by QCA) using any percutaneous method, without the occurrence of death, Myocardial Infarction (MI), or repeat revascularization of the target lesion during the hospital stay.
Time Frame: At procedure during hospital stay
Population: Intent to Treat
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 450 | 226
Percentage of participants | 97.3 | 98.7
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.407, Fisher Exact; Difference between event rates = -1.3, 95% CI 2-sided [-3.5 to 1.4]

6. Secondary Outcome: Percentage of Participants Who Experienced Target Lesion Revascularization (TLR)
Description: TLR is defined as any "clinically-driven" repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel. Clinically-driven revascularizations are those in which the patient has a positive functional study, ischemic electrocardiogram (ECG) changes at rest in a distribution consistent with the target vessel, or ischemic symptoms, and an in-lesion diameter stenosis 50 percent by QCA.
Time Frame: 12 months post-procedure
Population: Event specific adjusted ITT population: All randomized participants excluding those with follow-up less than 330 days and without documented events during the 360 days post procedure
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 429 | 216
Percentage of participants | 3.50 | 1.39
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.203, Fisher Exact; Difference between event rates = 2.11, 95% CI 2-sided [-0.84 to 4.48]

7. Secondary Outcome: Percentage of Participants Who Experienced Target Vessel Revascularization (TVR)
Description: TVR is defined as any "clinically driven" repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel. Clinically-driven revascularizations are those in which the patient has a positive functional study, ischemic ECG changes at rest in a distribution consistent with the target vessel, or ischemic symptoms, and an in-lesion diameter stenosis 50 percent by QCA.
Time Frame: 12 months post procedure
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 429 | 216
Percentage of participants | 5.13 | 2.78
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.22, Fisher Exact; Difference between event rates = 2.35, 95% CI 2-sided [-1.24 to 5.28]

8. Secondary Outcome: Percentage of Participants Who Experienced Target Vessel Failure (TVF)
Description: Target Vessel failure is defined as clinically-driven target lesion revascularization, target vessel myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel at 12 months post-procedure.
Time Frame: 12 months post procedure
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 429 | 216
Percentage of participants | 6.99 | 4.17
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.166, Fisher Exact; Difference between event rates = 2.83, 95% CI 2-sided [-1.28 to 6.26]

9. Secondary Outcome: Percentage of Participants Who Experienced Major Adverse Cardiac Events (MACE)
Description: MAJOR ADVERSE CARDIAC EVENTS (MACE) consists of death, myocardial infarction, emergent bypass surgery, and target lesion revascularization.
Time Frame: 12 months post procedure
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 429 | 216
Percentage of participants | 6.29 | 3.70
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.200, Fisher Exact; Difference between event rates = 2.59, 95% CI 2-sided [-1.35 to 5.85]

10. Secondary Outcome: Percentage of Participants Who Had Lesions of More Than 1 Vessel and Experienced Target Lesion Failure (TLF)
Description: A Target Lesion Failure is defined as clinically-driven target lesion revascularization, target vessel myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel at 12 months post-procedure.
Time Frame: 12 months post procedure
Population: All randomized participants with lesions of more than 1 vessel and were followed for 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 47 | 30
Percentage of participants | 14.89 | 3.33
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.140, Fisher Exact; Difference between event rates = 11.56, 95% CI 2-sided [-3.73 to 24.64]

11. Secondary Outcome: Percentage of Participants Who Had Diabetes and Experienced Target Lesion Failure (TLF)
Description: as for outcome 10
Time Frame: 12 months post procedure
Population: All randomized participants who had diabetes and were followed up for 12 months.
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 135 | 67
Percentage of participants | 6.67 | 1.49
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.170, Fisher Exact; Difference between event rates = 5.17, 95% CI 2-sided [-2.03 to 10.83]

12. Secondary Outcome: Percentage of Participants Who Experienced Bleeding Complications
Description: Bleeding complications include any bleeding events defined by THROMBOLYSIS IN MYOCARDIAL INFARCTION (TIMI), Global Strategies for Opening Occluded Coronary Arteries (GUSTO), and "Protocol" definitions.
Time Frame: 12 months post procedure
Population: All randomized participants who had 12 months follow-up and documented specific events
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 218
Percentage of participants | 13.08 | 12.84
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 1.0, Fisher Exact; Difference between event rates = 0.24, 95% CI 2-sided [-5.61 to 5.43]

13. Secondary Outcome: Percentage of Participants Who Died
Description: Death incidences include both Cardiac and non-cardiac death.
Time Frame: 12 months post procedure
Population: All randomized participants who had 12 months follow-up and documented specific events
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 0.70 | 0.46
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 1.0, Fisher Exact; Difference between event rates = 0.24, 95% CI 2-sided [-1.92 to 1.63]

14. Secondary Outcome: Percentage of Participants Who Experienced Any Myocardial Infarction (MI)
Description: Myocardial Infarction includes both Q-wave and WHO Non-Q Wave Myocardial Infarction events.
Time Frame: 12 months post procedure
Population: All randomized participants who had 12 months follow-up and documented specific events
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 2.80 | 2.31
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.801, Fisher Exact; Difference between event rates = 0.49, 95% CI 2-sided [-2.73 to 2.91]

15. Secondary Outcome: Percentage of Participants Who Experienced Stroke
Description: The stroke definition includes both hemorrhagic and non-hemorrhagic strokes.
Time Frame: 12 months post procedure
Population: All randomized participants who had 12 months follow-up and documented specific events
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 0.47 | 1.39
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.341, Fisher Exact; Difference between event rates = -0.92, 95% CI 2-sided [-3.56 to 0.60]

16. Secondary Outcome: Percentage of Participants Who Experienced Stent Thrombosis (Protocol Definition)
Description: Protocol defined Stent thrombosis include both Early and Late Thrombosis. Early thrombosis is defined as composite thirty-day ischemic endpoint including death, Q-wave MI, or subabrupt closure requiring revascularization. Late thrombosis is defined as myocardial infarction occurring > 30 days after the index procedure and attributable to the target vessel with angiographic documentation (site-reported or by qualitative coronary angiography) of thrombus or total occlusion at the target site and freedom from an interim revascularization of the target vessel.
Time Frame: 12 months post procedure
Population: Event specific adjusted ITT population: All randomized participants excluding those with follow-up less than 330 days and without documented specific events during the 360 days post procedure
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 0.47 | 0.46
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 1.00, Fisher Exact; Difference between event rates = 0.00, 95% CI 2-sided [-2.14 to 1.28]

17. Secondary Outcome: Percentage of Participants Who Experienced Stent Thrombosis (Academic Research Consortium (ARC) Definition)
Description: Academic Research Consortium (ARC) defines STENT THROMBOSIS as consisting of the following:
  1. DEFINITE - Angiographic or pathologic confirmation;
  2. PROBABLE - Any unexplained death within the first 30 days or Any MI (related to documented acute ischemia and without another obvious cause) in the territory of the stent;
  3. POSSIBLE - Any unexplained death > 30 days.
  ARC Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points.
Time Frame: 12 months post procedure
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 0.93 | 0.46
Statistical Analysis 1: Comparison: ELITE™ vs CYPHER®; Test type: Superiority or Other; p = 0.668, Fisher Exact; Difference between event rates = 0.47, 95% CI 2-sided [-1.72 to 1.96]

18. Secondary Outcome: Percentage of Participants Who Experienced Early Stent Thrombosis (Academic Research Consortium (ARC) Definition)
Description: Those ARC stent thromboses occurred between 0 and 30 days post-procedure are early stent thrombosis.
Time Frame: 0-30 days post-procedure
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 447 | 225
Percentage of participants | 0.22 | 0.00

19. Secondary Outcome: Percentage of Participants Who Experienced Late Stent Thrombosis (Academic Research Consortium (ARC) Definition)
Description: Those ARC stent thromboses occurred between 31 to 360 days post-procedure are late stent thrombosis.
Time Frame: 31-360 days post-procedure
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | ELITE™ | CYPHER®
Number analyzed (Participants) | 428 | 216
Percentage of participants | 0.7 | 0.46

ADVERSE EVENTS:
Arm/Group | ELITE™ | CYPHER®
Serious Adverse Events (participants affected / at risk) | 3/452 | 1/226
Other Adverse Events (participants affected / at risk) | 227/452 | 125/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELITE™ (N=452) | CYPHER® (N=226)
Death (Vascular disorders) | 3 (3) | 1 (1) — The deaths for the three patients were not MedDRA coded as "death" since these are based on site reported MedDRA coding to the underlying cause of death.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELITE™ (N=452) | CYPHER® (N=226)
Angina pectoris (Cardiac disorders) | 99 (99) | 64 (64)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 7 (7)
Bradycardia (Cardiac disorders) | 5 (5) | 3 (3)
Myocardial infarction (Cardiac disorders) | 21 (21) | 8 (8)
Catheter site haematoma (General disorders) | 11 (11) | 12 (12)
Catheter site haemorrhage (General disorders) | 21 (21) | 6 (6)
Catheter site pain (General disorders) | 5 (5) | 5 (5)
Non-cardiac chest pain (General disorders) | 7 (7) | 10 (10)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Hypersensitivity (Immune system disorders) | 6 (6) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Coronary revascularisation (Surgical and medical procedures) | 36 (36) | 14 (14)
Haemorrhage (Vascular disorders) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 12 (12) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 5 (5) | 2 (2)
Hypotension (Vascular disorders) | 9 (9) | 11 (11)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Artery dissection (Vascular disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor for business reasons. Hence the data was under powered for hypothesis testing. No definitive conclusions can be made from this data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days